CLINICAL TRIAL: NCT03339895
Title: Comparison of PVI-guided Fluid Management With Traditional Fluid Management in Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Sevim Cesur, DR, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: KOU KAEK 2015/99
Record Dates: First submitted 2017-01-30; First posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Fluid Overload
Keywords: COLORECTAL SURGERY; PVI GUIDED FLUID MANAGEMENT; GOAL DIRECTED THERAPY
MeSH Terms: conditions — Edema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pvı-guided (Experimental): pvı-guided(according to pvi value) fluid infused during whole procedure 2 ml/kg/h infusion during surgery
  Interventions: Other: pvı-guided
- traditional-guided (Experimental): 4-8 ml/kg/h infusion during surgery
  Interventions: Other: traditional-guided

INTERVENTIONS:
Other: pvı-guided — pvı- guided total amount of crystalloid volume of fluid infused during colorectal surgery pvı-guided(according to pvi value) fluid infused during whole procedure 2 ml/kg/h infusion during surgery If PVI value <%13 and if MAP>65mmHg continue with 2 ml/kg/h cristalloid infusion If PVI value <%13 and if MAP>65mmHg 5 mcg efedrin intravenous bolus till MAP>65 mmHg If PVI value >%13 and MAP>65 mmHg infuse 250 ml Gelofusine bolus up to PVI value lowers to %13 every 5 minute If PVI value >%13 and MAP <65 mmHg infuse 250 ml Gelofusine bolus and 5 mcg efedrin intravenous up to PVI value lowers to %13
  Arms: pvı-guided
Other: traditional-guided — traditional-guided total amount of crystalloid volume of fluid infused during colorectal surgery traditional-guided fluid infused during whole procedure 4-8 ml/kg/h infusion during surgery If MAP <65 mmHg or <30%of basal value, infuse 250 ml Gelofusine bolus and 5 mcg efedrin If MAP>65 mmHg no intervention
  Arms: traditional-guided

SUMMARY:
The first objective of this study was to compare the traditional fluid management (TFM) with PVI guided goal-directed fluid management (GDFM) in terms of controlled intraoperative fluid volume, surgical end-point fluid balance, blood lactate and serum creatinine levels. ASA I-II 70 patients included in this prospective study.

DETAILED DESCRIPTION:
Objectives: The first objective of our study was to compare the traditional fluid management (TFM) with PVI guided goal-directed fluid management (GDFM) in terms of controlled intraoperative fluid volume, surgical end-point fluid balance, blood lactate and serum creatinine levels. Our secondary purpose was to compare the effects of different fluid regimens on the return of bowel function and the duration of hospital stay. Methods: The study included 70 American Society of Anesthesiologists (ASA) grade I and II patients, aged above 18 and undergoing elective colorectal surgery. After premedication with 0.03 mg /kg i.v. midazolam, all patients were started an i.v. infusion of 500 mL 0.9 % NaCl until the end of anesthesia induction.

After the anesthesia induction, while 0.9 % NaCl at rate of 2 mL/kg/h was infused in PVI- guided GDFM group, a 250-mL bolus gelatin injection (Gelofusine®, Barun) was administered when PVI was higher than 13 % over 5 min. While 0.9 % NaCl at rate of 4- 8 mL/kg/h was infused in TFM group, a 250-ml bolus gelatin injection (Gelofusine®, Barun) was administered when the mean arterial blood pressure (MAP) decreased below 65 mmHg. In both groups, when MAP was still < 65 mmHg after fluid bolus infusion, 5 mg i.v. bolus ephedrine was administered. The data collected during intraoperative period, such as heart rate, MAP, arterial blood gas samples (Ph, arterial oxygen pressure (PaO2), arterial carbon dioxide pressure (PaCO2), HCO3 level, hemoglobin, blood lactate level) were recorded. Hemoglobin, Na, K, Cl, serum creatinine, blood lactate and serum albumin scores were measured preoperatively, and up to 24 hours postoperative.

In the first 24 hours after surgery, oliguria (<0.5 ml / kg urine output), need for blood transfusion and the time of first bowel movement (depending on the days after surgery), length of hospital stay were recorded.

ELIGIBILITY:
Inclusion Criteria:

* > 18 age
* elective colorectal suregry
* ASA 1-2

Exclusion Criteria:

* Chronic renal disease
* Ejection fraction < 30
* arthmia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-25 (Actual)

PRIMARY OUTCOMES:
FLUID MANAGEMENT | two hours
  total fluid given during colorectal surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sevim Cesur, MD, Principal Investigator — Specialist; Tülay Hoşten, MD, Study Director — Specialist

IPD SHARING:
Plan to Share IPD: No